CLINICAL TRIAL: NCT05752487
Title: Safety and Effectiveness Evaluation of the THERMOCOOL SMARTTOUCH SF Catheter With the TRUPULSE Generator for Treatment of Paroxysmal Atrial Fibrillation (PAF)
Brief Title: A Study For Treatment Of Paroxysmal Atrial Fibrillation (PAF) With The THERMOCOOL SMARTTOUCH SF Catheter and TRUPULSE Generator
Acronym: SmartfIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI202202; BWI202202 (Other: Biosense Webster, Inc.)
Record Dates: First submitted 2023-02-22; First posted 2023-03-02 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Pulsed Field (PF) /Radiofrequency (RF) Catheter ablation (Experimental): Participants with drug refractory, paroxysmal atrial fibrillation (PAF) who are candidates for catheter ablation will be enrolled with ablation system which uses THERMOCOOL SMARTTOUCH SF (STSF) catheter and TRUPULSE generator to deliver RF or PF energy during cardiac ablation procedures.
  Interventions: Device: Pulsed Field (PF) /Radiofrequency (RF) Catheter ablation

INTERVENTIONS:
Device: Pulsed Field (PF) /Radiofrequency (RF) Catheter ablation — Participants will undergo catheter ablation with the PF /RF ablation system consisting of the TRUPULSE Generator (delivers RF or PF energy through the study catheter) and the THERMOCOOL SMARTTOUCH SF (STSF) Catheter (indicated for use in catheter-based cardiac electrophysiological mapping (stimulating and recording) and, when used with a Generator, for cardiac ablation).

SUMMARY:
The purpose of this study is to demonstrate safety and effectiveness of the ablation system (THERMOCOOL SMARTTOUCH SF [STSF] catheter and TRUPULSE generator) when used for isolation of the atrial pulmonary veins (PVs) in treatment of participants with paroxysmal atrial fibrillation (PAF).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic paroxysmal atrial fibrillation (PAF) defined as atrial fibrillation (AF) that terminates spontaneously or with intervention within 7 days of onset. This PAF is considered to be symptomatic if symptoms related to AF are experienced by the participant
* Selected for AF ablation procedure by pulmonary vein isolation (PVI)
* Failed at least one antiarrhythmic drug (AAD) (class I to IV) as evidenced by recurrent symptomatic AF, or intolerable or contraindicated to the AAD
* Willing and capable of providing consent
* Able and willing to comply with all pre-, post- and follow-up testing and requirements.

Exclusion Criteria:

* Previously known AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause (example, documented obstructive sleep apnea, acute alcohol toxicity, morbid obesity {Body Mass Index greater than [>] 40 kilograms per meter square [kg/m²]}, renal insufficiency (with an estimated creatinine clearance less than [<] 30 milliliters [mL]/ minute [min]/1.73 meter square [m2] )
* Previous left atrium (LA) ablation or surgery
* Patients known to require ablation outside the pulmonary vein (PV) region (example, atrioventricular reentrant tachycardia, atrioventricular nodal reentry tachycardia, atrial tachycardia, ventricular tachycardia and wolff-parkinson-white)
* Previously diagnosed with persistent AF [greater than (>) 7 days in duration]
* Severe dilatation of the left atrium (LA) (Left anterior descending artery [LAD] >50mm antero-posterior diameter in case of Transthoracic Echocardiography [TTE])

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2024-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biosense Webster, Inc. Clinical Trial, Study Director — Biosense Webster, Inc.
Locations (9):
- Austria (2):
  - Medical University Graz, Graz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
- Belgium (4):
  - O L V Ziekenhuis, Aalst
  - AZ Sint-Jan, Bruges
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis, Hasselt
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Gentofte Hospital, Hellerup
- Vilnius University Hospital Santaros Clinics, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] De Potter T, Scherr D, Purerfellner H, Rackauskas G, Hansen J, Vijgen J, Phlips T, Knecht S, Szeplaki G, Van Herendael H, Kronborg MB, Berte B, Ruwald M, Kollias G, Lukac P, Tan T, Duytschaever M. Dual energy for pulmonary vein isolation using focal ablation technology integrated with a three-dimensional mapping system: SmartfIRE 12-month results. Europace. 2025 Sep 1;27(9):euaf174. doi: 10.1093/europace/euaf174. PMID 40796332
- [Derived] Duytschaever M, Rackauskas G, De Potter T, Hansen J, Knecht S, Phlips T, Vijgen J, Scherr D, Szeplaki G, Van Herendael H, Kronborg MB, Berte B, Purerfellner H, Lukac P. Dual energy for pulmonary vein isolation using dual-energy focal ablation technology integrated with a three-dimensional mapping system: SmartfIRE 3-month results. Europace. 2024 May 2;26(5):euae088. doi: 10.1093/europace/euae088. PMID 38696675

RESULTS

PARTICIPANT FLOW:
Groups:
- Pulsed Field (PF) /Radiofrequency (RF) Catheter Ablation: Participants with drug refractory, paroxysmal atrial fibrillation (PAF) who were candidates for catheter ablation were enrolled and treated with THERMOCOOL SMARTTOUCH SF (STSF) catheter and TRUPULSE generator to deliver radiofrequency (RF) or pulse field (PF) energy during cardiac ablation procedures .
Period: Overall Study
Arm/Group | Pulsed Field (PF) /Radiofrequency (RF) Catheter Ablation
Started | 149
Study Catheter Inserted | 140
Completed | 137
Not Completed | 12
Not completed — Enrolled, not treated | 9
Not completed — Study catheter inserted but did not undergo ablation | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Modified intention-to-treat (mITT) analysis set included all enrolled participants who met eligibility criteria and had insertion of the study catheter.
Arm/Group | Pulsed Field (PF) /Radiofrequency (RF) Catheter Ablation
Number analyzed (Participants) | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (7.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Race and Ethnicity were not collected from any participant. Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Primary Adverse Events (PAEs)
Description: Percentage of participants with PAEs (within 7 days following the ablation procedure) was reported. PAEs included the following adverse events atrio-esophageal fistula, pulmonary vein stenosis, device or procedure related death, (that occurred greater than 7 days and less than or equal to 90 days post-procedure), phrenic nerve paralysis (permanent), cardiac tamponade/perforation, stroke/cerebrovascular accident (CVA), major vascular access complication/bleeding, thromboembolism, myocardial infarction, transient ischemic attack (TIA), pericarditis, heart block, pulmonary edema (respiratory insufficiency), and vagal nerve injury/gastroparesis.
Time Frame: 90 days post-procedure on Day 1
Population: Modified intention-to-treat (mITT) analysis set included all enrolled participants who met eligibility criteria and had insertion of the study catheter. Here, 'N' (number of participants analyzed) refers to participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Pulsed Field (PF) /Radiofrequency (RF) Catheter Ablation
Number analyzed (Participants) | 137
percentage of participants
  Atrio-esophageal Fistula | 0.0
  Phrenic Nerve Paralysis (permanent) | 0.0
  Pulmonary Vein Stenosis | 1.5
  Cardiac Tamponade/perforation | 1.5
  Stroke/Cerebrovascular Accident (CVA) | 0.7
  Transient Ischemic Attack (TIA) | 0.0
  Major Vascular Access Complication / Bleeding | 0.0
  Thromboembolism | 0.0
  Myocardial Infarction | 0.0
  Pericarditis | 0.7
  Heart Block | 0.0
  Pulmonary Edema (Respiratory Insufficiency) | 0.0
  Vagal Nerve injury/Gastroparesis | 0.0
  Death (Device or procedure related) | 0.0

2. Primary Outcome: Percentage of Participants With Acute Procedural Success
Description: Percentage of participants with acute procedural success were reported. Procedural success was defined as electrical isolation of clinically relevant targeted pulmonary veins (PVs) (confirmed by entrance block) after adenosine/isoproterenol challenge at the end of the index ablation procedure.
Time Frame: Immediately post-procedure on Day 1
Population: The per protocol analysis set included enrolled eligible participants who had undergone ablation using PF and/or RF energy via the investigational ablation system per clinical investigational plan (CIP), were treated for the study-related arrythmia, and without major CIP deviation that effected the scientific integrity of the safety and effectiveness.
Measure: Number; unit: Percentage of participants
Arm/Group | Pulsed Field (PF) /Radiofrequency (RF) Catheter Ablation
Number analyzed (Participants) | 137
Percentage of participants | 100

3. Secondary Outcome: Percentage of Participants With Freedom From Documented (Symptomatic and Asymptomatic) Atrial Arrhythmia
Description: Percentage of participants with freedom from documented (symptomatic and asymptomatic) atrial arrhythmia episodes including atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL; unknown origin) episodes based on electrocardiographic data (greater than equal to [>=]30 seconds on arrhythmia monitoring device) were reported. Participants with an AF/AT/AFL (of unknown origin) episode that is >=30 seconds on arrhythmia monitoring device during the evaluation period were considered failures of this long-term effectiveness outcome measure. Acute procedural failure (that is, failure to achieve entrance block with the study device in any of the targeted pulmonary vein [PVs]) were also deemed a failure of this outcome measure. AFL of unknown origin was defined as all AFL except those cavotricuspid isthmus (CTI) dependent AFL as confirmed by 12-lead electrocardiogram (ECG) or entrainment maneuvers in an electrophysiology (EP) study.
Time Frame: Day 91 to Day 365
Population: The per protocol analysis set included enrolled eligible participants who had undergone ablation using PF and/or RF energy via the investigational ablation system per clinical investigational plan (CIP), were treated for the study-related arrythmia, and without major CIP deviation that effected the scientific integrity of the safety and effectiveness. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Pulsed Field (PF) /Radiofrequency (RF) Catheter Ablation
Number analyzed (Participants) | 134
Percentage of participants | 71.6

ADVERSE EVENTS:
Time Frame: From screening (Day -60) up to 12 months
Description: Safety data was analyzed based on all enrolled participants.
Arm/Group | Pulsed Field (PF) /Radiofrequency (RF) Catheter Ablation
All-Cause Mortality (participants affected / at risk) | 0/149
Serious Adverse Events (participants affected / at risk) | 23/149
Other Adverse Events (participants affected / at risk) | 90/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulsed Field (PF) /Radiofrequency (RF) Catheter Ablation (N=149)
Atrial flutter (Cardiac disorders) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 2 (2)
Diverticulitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hemianaesthesia (Nervous system disorders) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulsed Field (PF) /Radiofrequency (RF) Catheter Ablation (N=149)
Atrial tachycardia (Cardiac disorders) | 5 (6)
Palpitations (Cardiac disorders) | 4 (4)
Bradycardia (Cardiac disorders) | 3 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Chronotropic incompetence (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Encephalomalacia (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (3)
Amnesia (Nervous system disorders) | 1 (2)
Aura (Nervous system disorders) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Ophthalmic migraine (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Chest pain (General disorders) | 4 (4)
Swelling (General disorders) | 2 (2)
Exercise tolerance decreased (General disorders) | 2 (2)
Medical device site reaction (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 7 (7)
Haemorrhage (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 3 (3)
COVID-19 (Infections and infestations) | 6 (6)
Bronchitis (Infections and infestations) | 2 (2)
Candida infection (Infections and infestations) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Atrial flutter (Cardiac disorders) | 16 (16)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Laryngeal injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Pharyngeal injury (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Heart rate increased (Investigations) | 2 (2)
Haematuria (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Puncture site haemorrhage (General disorders) | 4 (4)
Puncture site pain (General disorders) | 3 (3)
Cystitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Nasal vestibulitis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1)
Anosmia (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Rectal lesion (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Glaucoma (Eye disorders) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Spirometry (Investigations) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Hereditary haemochromatosis (Congenital, familial and genetic disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT05752487/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT05752487/SAP_001.pdf